CLINICAL TRIAL: NCT02180191
Title: Comparison of Gut Microbiota in Obese, Diabetic and Healthy Control Individuals
Brief Title: Gut Microbiota in Obesity and Diabetes
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Yalcin Basaran, MD, Gulhane School of Medicine
Other Study IDs: GSM-2012/48; GSM-2012 (Other: Gulhane School of Medicine-2012)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Gut microbiota
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Obesity: 27 obese individuals (20 men and 7 women with mean BMI: 39.98±5.56 kg/m2)
  Interventions: Other: Comparison of the gut microbiota composition
- Diabetes: 26 patients with newly diagnosed type 2 diabetes (18 men and 8 women with mean BMI: 28.63±5.08 kg/m2)
  Interventions: Other: Comparison of the gut microbiota composition
- Control: Healthy control subjects (22 men and 6 women with mean BMI: 23.02±1.70 kg/m2)
  Interventions: Other: Comparison of the gut microbiota composition

INTERVENTIONS:
Other: Comparison of the gut microbiota composition

SUMMARY:
An altered gut microbiota composition has recently been linked to obesity and diabetes. The principal aim of this study was to investigate and compare the gut microbiota composition of obese, diabetic and control individuals. Then, associations between analyzed gut microbial concentrations and clinical-biochemical blood parameters were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with obesity or newly diagnosed type 2 diabetes
* 18 years to 65 years of age

Exclusion Criteria:

* Any chronic disease (other than obesity and diabetes)
* Alcohol consumption/smoking
* Pregnancy/breastfeeding
* The use of antibiotics, pro-prebiotics within 3 months
* <18 years or >65 years
* History of intestinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The comparison of the gut microbiota composition | 9 months
  The gut microbiota composition of obese, diabetic and control individuals was analyzed by quantitative real-time PCR (qRT-PCR)

SECONDARY OUTCOMES:
The relationship between metabolic parameters and the gut microbiota composition | 9 months
  A multivariate linear regression analysis was performed in order to test associations between the gut microbiota composition and metabolic variables of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Metabolism, Gulhane School of Medicine, Ankara, Turkey (Türkiye)